CLINICAL TRIAL: NCT03260881
Title: Effects of Liraglutide on Epicardial Fat Pro-Inflammatory Genes in Type 2 Diabetes and Coronary Artery Disease
Brief Title: Liraglutide Effects on Epicardial Fat Inflammatory Genes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Gianluca Iacobellis, Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20170684
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Type2 Diabetes; Coronary Artery Disease
Keywords: Epicardial Fat
MeSH Terms: conditions — Coronary Artery Disease | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: Double-blind, parallel group, placebo controlled study.
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind, parallel group, placebo controlled study. The method of allocation generation will be a computerized random-number generator. The sequence will be generated by the process of restricted randomization. Computer-based randomization process will be managed by the UM Research pharmacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-group (Active Comparator): • L-group will be started on liraglutide. Liraglutide will be started and administered for from a minimum of 4 weeks up to 12 weeks prior to CABG with a starting dose of 0.6 mg (after a least one week) and subsequent increments to 1.2 mg (after a least one week) and to 1.8 mg (after at least a week on 1.2 mg). The dose of 1.8 mg daily will be maintained until the end of the 12-week study. Other and current diabetes treatment will be continued
  Interventions: Drug: Liraglutide Pen Injector [Victoza]
- D-group (Placebo Comparator): placebo will be administered in addition to current treatment prior to the CABG with a starting dose of 0.6 mg (after a least one week) and subsequent increments to 1.2 mg (after a least one week) and to 1.8 mg (after at least a week on 1.2 mg). D-group will be started on a supervised low calorie diet (LCD) to achieve approximately 5% of weight loss after from a minimum of 4 weeks up to 12 weeks.
  Interventions: Drug: matching liraglutide-placebo pre-filled pens

INTERVENTIONS:
Drug: Liraglutide Pen Injector [Victoza] — Study subjects will be randomized in two groups of 20 patients to receive additional liraglutide, (L-group) or to remain on current treatment or placebo (D-group).
  Arms: L-group
Drug: matching liraglutide-placebo pre-filled pens — Study subjects will be randomized in two groups of 20 patients to receive additional liraglutide, (L-group) or to remain on current treatment or placebo (D-group).
  Arms: D-group

SUMMARY:
Epicardial adipose tissue (EAT) is the visceral fat of the heart. EAT could locally affect the coronary arteries through local secretion of pro-inflammatory cytokines. EAT plays a role in the development of the coronary artery disease (CAD). EAT is a highly enriched with genes involved in inflammation. Given its rapid metabolism and simple measurability, as first developed by Iacobellis, EAT serves as target for medications targeting the fat. Glucagon-like peptide-1 agonists (GLP-1A) are anti-diabetic medications with recently suggested cardio-protective properties. Liraglutide, a GLP-1A, has recently shown to reduce the cardiovascular risk. Iacobellis'group found that EAT thickness decreased by an unprecedented 36% after 12 weeks of treatment with liraglutide. Remarkably, Iacobellis'group found for the first time that human EAT express GLP-1 Receptor (GLP-1R). GLP-1A effects may be therefore visceral fat specific and target EAT. Based on these preliminary data, we hypothesize that treatment with liraglutide will significantly and rapidly reduce EAT inflammation. Decreased EAT inflammation can reduce the burden of the coronary plaques. We will test our hypothesis in a 12-week randomized, double-blind, placebo-controlled, interventional study in 40 patients with type 2 diabetes mellitus (T2DM), and CAD, with an acceptable glycemic control on their current diabetes regimen who require elective coronary artery bypass graft (CABG) regardless of their participation in the study. A minimum time frame of 3-week treatment will be considered to detect significant changes in the study endpoints. Inclusion criteria for body fat markers will rule out the confounding effect of different body fast distribution at baseline. Study subjects will be randomized in two groups of 20 patients to receive additional liraglutide or to remain on current treatment/ placebo prior to cardiac surgery. CAD subjects not allocated to liraglutide will be started on a supervised low-calorie diet (LCD) to achieve approximately 5% of weight loss after from a minimum of 3 weeks up to 12 weeks to avoid the confounding effect of weight loss on the study outcomes. Fat samples will be collected during cardiac surgery after up to 12 weeks of treatment either with liraglutide or placebo and processed for analysis of mRNA and protein expression of EAT and SAT inflammatory genes such as Tumor Necrosis Factor-alpha (TNF-α) and Interleukin 6 (IL-6), and GLP-1R.

ELIGIBILITY:
Inclusion Criteria:

* T2DM as defined by American Diabetes Association (ADA) criteria
* Adult patients with T2DM who are indicated to receive liraglutide, not as first-line therapy, in addition to diet and exercise to improve glycemic control
* Hemoglobin A1c (HbA1c) ≤ 9%
* Age ≥ 18 years old
* Body mass index (BMI) ≥ 27 Kg/m2 and/or waist circumference ≥ 102 cm (40 inches) in men and 88 cm (35 inches) in women, respectively.
* Clinically and angiographically stable CAD who requires CABG as part of the standard medical care, as CAD does not represent a contraindication for using liraglutide. The stability of the CAD further warranties that study patients will not be exposed to higher risk by using liraglutide

Exclusion Criteria:

* Patients with a personal or family history of medullary thyroid carcinoma or patients with Multiple Endocrine Neoplasia syndrome type 2
* Patients with a prior serious hypersensitivity reaction to liraglutide
* Other contra-indications to liraglutide in accordance with risks and safety information included in the latest updated prescribing information
* Type 1 diabetes, as defined by ADA criteria
* Current use of other GLP-1A, dipeptidyl peptidase 4 (DPP4) or Sodium Glucose transporters 2 (SGLT2) inhibitors, thiazolidinediones (TZDs), pramlintide and fixed prandial insulin.
* Patients with unstable CAD, assessed by the Cardiology team and defined as new onset angina, rest angina, rapidly increasing or crescendo angina
* History of diabetic ketoacidosis, pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy; acute or chronic infective diseases, cancer or chemotherapy, history of pulmonary, renal or liver diseases, and drug abuse
* Patients with chronic and acute inflammatory conditions such as sepsis, rheumatoid arthritis, ectopic dermatitis, asthma, ulcerative colitis.
* Current use of systemic corticosteroids in the 3 months prior this study.
* Pregnant or breast-feeding women
* Females of childbearing potential who are not using adequate contraceptive methods (as required by local law or practice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Iacobellis, MD PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited among the outpatient population who routinely referred to the University of Miami, Division of Cardiothoracic Surgery, and/or the Division and/or Division of Endocrinology, Diabetes and Metabolism outpatient clinics who required elective coronary artery bypass graft (CABG) surgery regardless of their participation in the study during COVID-19 pandemic
Groups:
- Study Group: Study group was started on liraglutide in addition to current standard treatment for diabetes and CAD for a minimum of 4 weeks up to 12 weeks prior to CABG with a starting dose of 0.6 mg (after a least one week) and subsequent increments to 1.2 mg (after a least one week) and to 1.8 mg (after at least a week on 1.2 mg), or maximum tolerated dose (MTD).
- Control Group: Control group received placebo pens in addition to current treatment for a minimum of 4 weeks up to 12 weeks prior to the CABG with a starting dose of 0.6 mg (after a least one week) and subsequent increments to 1.2 mg (after a least one week) and to 1.8 mg (after at least a week on 1.2 mg). Patients continued placebo up to the day before CABG
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (7) | 65 (11) | 64.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 15 | 15 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.7 (6.1) | 32.1 (6.8) | 32.4 (6.4)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: %HbA1C] | 6.9 (1.1) | 7.2 (1.3) | 7 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: EAT Inflammation
Description: EAT adipogenesis and inflammation as measured by miRNA expression (miR16-miR155-miR181a), from peri-coronary EAT samples collected during CABG after up to 12 weeks of treatment with either liraglutide or placebo. Tumor Necrosis Factor (TNF)-Alpha and Interleukin (IL)-6 gene expression were also measured in a subsample of peri-coronary EAT samples. miRNA and gene expression will be expressed as cycle threshold (ct) units. The PCR ct (cycle threshold) value refers to the number of cycles needed to replicate enough RNA to be detected.
Time Frame: Up to 12 weeks
Population: EAT fat samples could not be collected in 8 patients (5 in the liraglutide group and 3 in the placebo group) due to surgical circumstances and surgeon's decision during the CABG and in 2 patients (1 in the liraglutide and 1 in the placebo group) who eventually decided not to have surgery despite the clinical indications.
Measure: Median (Standard Deviation); unit: ct (cycle threshold)
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 13 | 15
ct (cycle threshold)
  miR16 | 0.70 (0.60) | 1.4 (2.3)
  miR155 | 0.39 (0.42) | 0.25 (0.43)
  miR181-a | 0.32 (0.42) | 0.25 (0.43)
  IL6: number analyzed (Participants) | 5 | 5
  IL6 | 0.8 (0.16) | 0.5 (0.14)
  TNF-a: number analyzed (Participants) | 5 | 5
  TNF-a | 0.57 (0.14) | 0.12 (0.05)

2. Secondary Outcome: EAT Thickness
Description: Change from baseline in EAT thickness as measured via ultrasound in mm
Time Frame: Baseline and up to 12 weeks
Population: EAT thickness ultrasound measurement could not be performed after the CABG due to COVID-19 hospital restrictions
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 19 | 19
mm | 11.8 (2.1) | 10 (2)

3. Secondary Outcome: SAT Inflammation
Description: SAT adipogenesis and inflammation as measured by miRNA expression (miR16-miR155-miR181a), from SAT samples collected during CABG after up to 12 weeks of treatment with either liraglutide or placebo. miRNA will be expressed as cycle threshold (ct) units. The PCR ct (cycle threshold) value refers to the number of cycles needed to replicate enough RNA to be detected.
Time Frame: Up to 12 weeks
Population: Fat samples could not be collected in 8 patients (5 in the liraglutide group and 3 in the placebo group) due to surgical circumstances and surgeon's decision during the CABG and in 2 patients (1 in the liraglutide and 1 in the placebo group) who eventually decided not to have surgery despite the clinical indications.
Measure: Median (Standard Deviation); unit: ct (cycle threshold)
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 13 | 15
ct (cycle threshold)
  miR16 | 0.08 (0.11) | 0.17 (0.36)
  miR155 | 0.06 (0.11) | 0.04 (0.07)
  miR181a | 0.12 (0.24) | 0.07 (0.16)

4. Secondary Outcome: Epicardial Adipose Tissue Glucagon Like 1 Receptor (EAT-GLP-1R)
Description: Gene expression of receptors or GLP-1 within EAT, expressed as cycle threshold (ct) units. The PCT Ct (cycle threshold) value refers to the number of cycles needed to replicate enough RNA to be detected
Time Frame: Up to 12 weeks
Population: Data was not collected due to due to technical difficulties and decision of the cardiac surgeon during the CABG surgery.
Arm/Group | L-group | D-group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: patients were followed up to 12 weeks from enrollment to the day of the CABG surgery
Arm/Group | Study Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 6/19 | 2/19
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Study Group (N=19) | Control Group (N=19)
nausea (Gastrointestinal disorders) | 6 | 2
abdominal distention (Gastrointestinal disorders) | 6 | 2

LIMITATIONS AND CAVEATS:
Overall, the study was greatly affected by the COVID-19 pandemic. Enrollment, clinical assessment, surgery schedule, fat sample collection were all impacted by COVID-19. Fat samples could not be collected or analyzed in all patients due to COVID-19 restrictions and surgical decisions during the standard of care CABG. Ultrasound EAT thickness could not be measured after the CABG due to COVID-9 restrictions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT03260881/Prot_SAP_000.pdf